CLINICAL TRIAL: NCT04746560
Title: Evaluation of the Diagnostic Performances of the TEG 6s® Hemostasis Device and Its Platelet Mapping® Cartridge for Perioperative Monitoring of Platelet Function During Cardiopulmonary Bypass for Cardiac Surgery
Brief Title: TEG 6s® for Perioperative Monitoring of Platelet Function During Cardiopulmonary Bypass for Cardiac Surgery
Acronym: TEG-PM
Status: Terminated | Type: Observational
Why Stopped: Haemonetics, the company that manages the TEG device, has given a negative answer as to the continuation of the study. For technical and internal reasons, they will take over the device.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201216
Record Dates: First submitted 2020-12-11; First posted 2021-02-10 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-09

CONDITIONS: Cardiopulmonary Bypass
Keywords: Cardiopulmonary bypass; Cardiac Surgery; Platelet function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TEG®6S device with its Platelet mapping® cartridge — Platelet function monitoring using the TEG®6S device with its Platelet mapping® cartridge

SUMMARY:
Excessive bleeding is common during cardiopulmonary bypass (CPB) for cardiac surgery. This may result from the systemic activation of the coagulation pathway and the acquired platelet dysfunction during the procedure. This study aims to compare the diagnostic performances of the TEG®6S device and its Platelet mapping® cartridge to those of the "gold standard" tests (light transmittance aggregometry and Multiplate®) for platelet function monitoring in patients undergoing CPB for cardiac surgery.

DETAILED DESCRIPTION:
Excessive bleeding is common during cardiopulmonary bypass (CPB) for cardiac surgery. This may result from the systemic activation of the coagulation pathway and the acquired platelet dysfunction during the procedure. This study aims to compare the diagnostic performances of the TEG®6S device and its Platelet mapping® cartridge to those of the "gold standard" tests (light transmittance aggregometry and Multiplate®) for platelet function monitoring in patients undergoing CPB for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo cardiopulmonary bypass
* Informed consent

Exclusion Criteria:

* Age <18 years
* Pregnant women
* Emergency surgery
* Cardiac surgery without CPB
* thrombocytopenia <100000/mmm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major persons operated on for cardiac surgery under extracorporeal circulation
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping cartridge with that of the reference tests used in the hematology laboratory for the evaluation of platelet function | 6 hours after inclusion
  Comparison of the results of reference tests used in the hematology laboratory for the evaluation of platelet function such as platelet aggregation in photometry (ADP, arachidonic acid, TRAP),with the results of the TEG® Platelet mapping® cartridge (MA fibrin, MA-ADP, MA-AA) obtained at the different pre, per and post-extracorporeal circulation sampling times
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping cartridge with that of the reference tests used in the hematology laboratory for the evaluation of platelet function | 6 hours after inclusion
  Comparison of the results of reference tests used in the hematology laboratory for the evaluation of platelet function such as the results of total blood aggregometry by impedance (Multiplate®: TRAPtest, ASPItest and ADPtest), with the results of the TEG® Platelet mapping® cartridge (MA fibrin, MA-ADP, MA-AA) obtained at the different pre, per and post-extracorporeal circulation sampling times

SECONDARY OUTCOMES:
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding. | 24 hours after inclusion
  Compare results obtained at different sampling times (pre, per and post-extracorporeal circulation) of the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding, using: ・ The results of platelet aggregation in photometry (ADP, arachidonic acid, TRAP)
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding. | 24 hours after inclusion
  Compare results obtained at different sampling times (pre, per and post-extracorporeal circulation) of the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding, using The results of total blood aggregometry by impedance (Multiplate®: TRAPtest, ASPItest and ADPtest)
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding. | 24 hours after inclusion
  Compare results obtained at different sampling times (pre, per and post-extracorporeal circulation) of the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding, using TEG® Platelet mapping® cartridge results (MA fibrin, MA-ADP, MA-AA)
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding. | 24 hours after inclusion
  Compare results obtained at different sampling times (pre, per and post-extracorporeal circulation) of the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding, using Global Haemostasis® cartridge results (R and K times, angle, amplitudes MA, A30 and A60) obtained at different sampling times
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding. | 24 hours after inclusion
  Compare results obtained at different sampling times (pre, per and post-extracorporeal circulation) of the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding, using Number and type of blood products transfused at the 24th hour after surgery
Compare the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding. | 24 hours after inclusion
  Compare results obtained at different sampling times (pre, per and post-extracorporeal circulation) of the diagnostic performance of the TEG®6S device and its Platelet mapping® cartridge with the reference tests used in the hematology laboratory for the prediction of the risk of post-cardiopulmonary bypass bleeding, using
  ・ The amount of bleeding in the drains at the 24th hour after surgery
Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass | 24 hours after inclusion
  Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass by statistical analysis of: ・ The results of platelet aggregation in photometry (ADP, arachidonic acid, TRAP)
Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass | 24 hours after inclusion
  Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass by statistical analysis of: ・ The results of total blood aggregometry by impedance (Multiplate®: TRAPtest, ASPItest and ADPtest)
Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass | 24 hours after inclusion
  Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass by statistical analysis of: ・ TEG® Platelet mapping® cartridge results (MA fibrin, MA-ADP, MA-AA)
Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass | 24 hours after inclusion
  Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass by statistical analysis of: ・ Global Haemostasis® cartridge results (R and K times, angle, amplitudes MA, A30 and A60) ; obtained at different sampling times
Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass | 24 hours after inclusion
  Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass by statistical analysis of: ・ Number and type of blood products transfused at the 24th hour after surgery
Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass | 24 hours after inclusion
  Evaluate the diagnostic performance of the TEG®6S device and its Global Haemostasis® cartridge in predicting the risk of bleeding at the end of cardiopulmonary bypass by statistical analysis of: ・ The amount of bleeding in the drains at the 24th hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Adrien BOUGLE, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Ahmed ABBES, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département d'Anesthésie-Réanimation,Hopital Pitié Salpêtrière, Paris, France